CLINICAL TRIAL: NCT05355129
Title: A Phase I, Randomized, Double-blind, Placebo-controlled, Ascending Single Dose and Multiple Dose Study of TT-00920 in Healthy Subjects
Brief Title: A Phase 1 Study of TT-00920 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TransThera Sciences (Nanjing), Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: TT00920CN02
Record Dates: First submitted 2022-04-05; First posted 2022-05-02 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Dose 1 (Experimental): low dose
  Interventions: Drug: TT-00920
- Dose 2 (Experimental): Middle dose
  Interventions: Drug: TT-00920
- Dose 3 (Experimental): High dose
  Interventions: Drug: TT-00920
- Placebo (Placebo Comparator)
  Interventions: Drug: TT-00920 Placebo

INTERVENTIONS:
Drug: TT-00920 — Tablets
  Arms: Dose 1; Dose 2; Dose 3
Drug: TT-00920 Placebo — Tablets
  Arms: Placebo

SUMMARY:
This is a double-blind, randomized, placebo-controlled, ascending single dose and multiple dose escalation study of TT-00920 in healthy subjects.

DETAILED DESCRIPTION:
This is a double-blind, randomized, placebo-controlled, ascending single dose and multiple dose escalation study of TT-00920 in healthy subjects. Each dosing cohort will comprise of 10 randomized subjects. Subjects received a single dose of TT-00920/ placebo during a single dose period, followed by a 3-10 day washout period, and then entered a 7-day multiple dose period, in which subjects received TT-00920/ placebo three times daily (TID) for days 1-6 and a single dose on day 7. The study will consist of a Screening Period, an In-house Period and a Follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained
* Age ≥ 18.0 years and ≤ 55.0 years, male or female
* BMI between 18.0 and 30.0 kg/m2, inclusive, and male weighs at least 50.0 kg and female weighs at least 45.0 kg

Exclusion Criteria:

* Known hypersensitivity or allergy to lactose
* Vaccination with any live vaccine, or vaccination employing an mRNA platform within 28 days and/or vaccination with any inactivated vaccine within 7 days of study drug administration
* Impaired cardiac function including clinically significant arrhythmias or clinically significant abnormality
* Subject with a history of severe visual diseases; or visual changes
* Subject is unable to complete this study for other reasons

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-11-03 (Actual); Primary Completion 2022-06-06 (Actual); Study Completion 2022-06-06 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Who Experience at Least One Treatment-emergent Adverse Event (TEAE) as assessed by Investigator | 20 days
  An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. A TEAE is defined as an adverse event that occurred or worsened after receiving study drug.
Percentage of Participants With Clinically relevant changes in vital signs | 20 days
  Vital signs include temperature, respiratory rate, blood pressure and pulse
Percentage of Participants With Clinically relevant changes in clinical laboratory tests | 20 days
  Safety laboratory tests includes hematology, coagulation, serum chemistries, and urinalysis.
Percentage of Participants With Clinically relevant changes in Electrocardiogram (ECG) | 20 days
  A standard 12-lead ECG was performed.

SECONDARY OUTCOMES:
Derived multiple dose PK parameters | 20 days
  AUC0 t, ss
Derived multiple dose PK parameters | 20 days
  Cmax, ss
Derived multiple dose PK parameters | 20 days
  tmax, ss
Derived multiple dose PK parameters | 20 days
  Rac
Derived multiple dose PK parameters | 20 days
  Cav
Derived multiple dose PK parameters | 20 days
  CL/F, ss
Derived single dose PK parameters | 20 days
  AUC0 t
Derived single dose PK parameters | 20 days
  Cmax
Derived single dose PK parameters | 20 days
  tmax

OTHER OUTCOMES:
TT-00920 metabolites as compared to baseline | 20 days
  AUC of observed drug-related material in plasma to determine the presence of any metabolite >10%
Change in Biomarkers From Baseline to Day 7: cGMP (Pmol/mL) | 20 days
  cGMP: cyclic guanosine monophosphate
Percentage of Subjects With an Actionable Genotype, Defined as the Presence of Any Mutation(s) That is (Are) Used to Guide a Drug/Dose Modification | 20 days
  An actionable genotype is defined as the presence of at least one mutation that is used to guide a drug/dose modification
Urine PK parameters | 20 days
  Aet
Urine PK parameters Feurine% | 20 days
  Feurine%: Fraction of drug excreted in urine

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China